CLINICAL TRIAL: NCT04434833
Title: A Single-cell Transcriptome Study in Patients With Non-Hodgkin's Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, First Deputy Director of Shanghai Institute of Hematology, Ruijin Hospital
Other Study IDs: NHL-scRNA
Record Dates: First submitted 2020-05-20; First posted 2020-06-17 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Extra nodal diseases: Patients with both lymph node and extra nodal involvement.
- Target drugs: Patients enrolled in clinical trials of novel target drugs.
- Relapse: Patients with high risk of relapse.

SUMMARY:
Using single-cell RNA sequencing, this study will explore the heterogeneity of lymphoma inside and outside the lymph node, identify tumor specific molecular markers and cell subgroups, explore the differences in tumor microenvironment composition, and provide a basis for diagnosis and precision treatment.

DETAILED DESCRIPTION:
In recent decades, the incidence of lymphoma has been increasing year by year in the world. Non-Hodgkin lymphoma accounts for about 90% of lymphoma, of which the classification is complex and the efficacy is poor compared to Hodgkin's lymphoma. Non-Hodgkin's lymphoma is often associated with the extra nodal involvement, and according to literature, extra nodal lymphoma accounts for 1/3 to 1/2 of all non-Hodgkin lymphomas. Compared with non-Hodgkin's lymphoma without extra nodal involvement, the prognosis of lymphoma with extra nodal involvement was relatively poor. The recurrence rate was higher, and its incidence, histology type, clinical staging and so on all had their own characteristics.

Tumor cells depend to some extent on the interaction with non-tumor cells and matrix components of the tumor microenvironment to maintain survival and proliferation. In addition, the non tumor cells and matrix components can mediate immunosuppressive action to promote tumor escape from immunosurveillance, resulting in disease progression. At the same time, more and more data show that the tumor microenvironment plays a key role in the development of tumor resistance. The cellular composition and spatial properties of the tumor microenvironment show significant heterogeneity, depending on a number of factors, including subtypes of lymphomas and extra nodal sites of lymphomas. Studying the tumor microenvironment will provide rationale for more precise target therapy. Through single-cell RNA sequencing, this study hopes to identify the heterogeneity of nodal and extra nodal lymphoma cells, to understand the differences in tumor microenvironment, and to provide a basis for diagnosis and precision treatment.

There are new target drugs for different antigen targets. But patients may not be sensitive to a certain drug, and the drug is often expensive, resulting in increased financial burden on patients without efficacy. Therefore, the research for biomarkers to predict patient efficacy and prognosis is particularly important.

The treatment efficacy of patients with relapsed lymphoma is often not good, so the prediction and treatment of patients with high-risk of relapsing is a clinical significant problem. On the basis of single-cell transcriptomics, this study hopes to find biomarkers for predicting the relapse of lymphoma and provide new ideas for clinical diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathological confirmed diagnosis of non-Hodgkin's lymphomas.
* Patients with both lymph node and extra nodal involvement, or patients at high risk of relapse, or patients receiving a novel target drug treatment.

Min Age: 14 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The tissue puncture specimens patients with both lymph node and extra nodal involvement, or patients at high risk of relapse, or patients receiving a novel target drug treatment will be obtained and restored for single-cell RNA sequencing.
  The clinical significance of single-cell RNA sequencing results will be explained combined with the clinical data provided by Ruijin Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Extra nodal involvement | At enrollment
  Clinical diagnosis of lymphoma invasion in extra nodal organs with or without pathological confirmation
Complete response rate | After 6 cycles of treatment (each cycle 21 to 28 days)
Overall response rate | After 6 cycles of treatment (each cycle 21 to 28 days)
Relapse | From the achievement of complete response to study completion, an average of 2 years
  Clinical diagnosis of emergence of new lymphoma lesion with or without pathology confirmation

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ruijin Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided